CLINICAL TRIAL: NCT02652247
Title: Serial, Non-invasive Molecular Analysis of Exhaled Breath Condensate to Define the Pulmonary Flora in Critically Injured, Ventilated Adults: The Clinical Trial
Brief Title: Serial, Non-invasive Analysis of Exhaled Breath Condensate in Ventilated Trauma Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: We did not have the funding to complete the study enrollment.
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Wonder Drake, Professor, Vanderbilt University Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 151194; 1R01GM115353-01 (NIH)
Record Dates: First submitted 2016-01-07; First posted 2016-01-11 (Estimated); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Ventilator Associated Pneumonia (VAP)
Keywords: trauma; ventilator; surgical ICU
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- ventilated trauma patients with pneumonia (Experimental): ventilated trauma patients with pneumonia
  Interventions: Procedure: molecular analysis of exhaled breath condensate; Procedure: molecular analysis of mini-bronchoalveolar lavage (BAL) aspirate; Procedure: molecular analysis of bronchoalveolar lavage (BAL) aspirate
- ventilated trauma patients without pneumonia (Experimental): ventilated trauma patients without pneumonia
  Interventions: Procedure: molecular analysis of exhaled breath condensate; Procedure: molecular analysis of mini-bronchoalveolar lavage (BAL) aspirate
- ventilated surgical ICU patients with pneumonia (Experimental): ventilated surgical ICU patients with pneumonia
  Interventions: Procedure: molecular analysis of exhaled breath condensate; Procedure: molecular analysis of mini-bronchoalveolar lavage (BAL) aspirate; Procedure: molecular analysis of bronchoalveolar lavage (BAL) aspirate
- ventilated surgical ICU patients without pneumonia (Experimental): ventilated surgical ICU patients without pneumonia
  Interventions: Procedure: molecular analysis of exhaled breath condensate; Procedure: molecular analysis of mini-bronchoalveolar lavage (BAL) aspirate

INTERVENTIONS:
Procedure: molecular analysis of exhaled breath condensate
Procedure: molecular analysis of mini-bronchoalveolar lavage (BAL) aspirate
Procedure: molecular analysis of bronchoalveolar lavage (BAL) aspirate
  Arms: ventilated surgical ICU patients with pneumonia; ventilated trauma patients with pneumonia

SUMMARY:
To determine if the analysis of exhaled breath condensate correlates with the development & resolution of pneumonia.

DETAILED DESCRIPTION:
This proposal investigates the utility of exhaled breath condensate fluid (EBCF) collected from heat moisture exchange (HME) filters connected to patient's endotracheal tubes for early, non-invasive detection of ventilator-associated pneumonia (VAP) in critically ill or injured ICU patients. The development of pneumonia during mechanical ventilation is the most common healthcare-associated infection in severely injured patients, accounting for substantial morbidity, excess ICU and hospital stay, additional cost and increased mortality.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Admitted to the Vanderbilt Trauma (TICU) and Surgical Intensive Care Units (SICU)
* Mechanically ventilated for ≥2 successive days (without planned extubation within 24 hours of enrollment)

Exclusion Criteria:

* Less than 18 years of age
* Expected survival less than 24 hours
* Anticipated extubation within 24 hours of enrollment
* Conditions limiting the subject's ability to tolerate collection of lavage specimens, including: FIO2 > 80%; PEEP > 16 cmH2O; Intracranial pressure >20 cmH2O; Tracheal or mucosal bleeding; Platelet count < 20,000 cells/uL; INR > 2.0
* Known prisoners
* Pneumonia diagnosis at the time of ICU admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2016-01; Primary Completion 2022-06 (Actual); Study Completion 2022-06 (Actual)

PRIMARY OUTCOMES:
The number of patients with a positive association between the exhaled breath condensate fluid and BAL fluid in in patients suspected of pneumonia. | enrollment to hospital day 15
  To determine the association between the microbial community in both EBCF specimens and bronchoalveolar lavage fluid (BALF) samples in critically ill and injured, mechanically ventilated patients suspected of VAP.
The per cent of positive correlation for the development & resolution of pneumonia based on changes in bacteria found in the exhaled breath condensate. | enrollment to hospital day 15
  To develop a robust predictive model for the development of VAP and its resolution based on changes in the microbial community in EBCF collected over the course of ventilation.

CONTACTS AND LOCATIONS:
Overall Officials: Addison K May, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No